CLINICAL TRIAL: NCT03992833
Title: Methods of Computed Tomography Screening and Management of Lung Cancer in Tianjin: A Population-based Cohort Study
Brief Title: Methods of Computed Tomography Screening and Management of Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: University Medical Center Groningen (Other); Shanghai Changzheng Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016YFE0103000
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Lung Neoplasms; Computed Tomography; Mass Screening; Lung Nodules
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung cancer screening (Experimental): Participants will undergo a chest CT scan in the Department of Radiology at Tianjin Cancer Hospital. All scans will be performed using the same CT system: Definition AS. Two readings of the images will be performed. In the first image reading, the CT images will be read by specially trained Chinese resident radiologist and checked by one of two senior Chinese radiologists. Lung Cancer Screening (version 2. 2018) Guidelines of the National Comprehensive Cancer Network (NCCN) will be used for the management of lung nodules. This guideline recommends management of lung nodules based on diameter. In the second reading, a semi-automated volumetry software will be used to measure the volume and evaluate the other parameters of lung nodules.
  At baseline and one year after baseline, data about general characteristics, risk factors of lung cancer, and health status of the participants will be collected.
  Interventions: Other: lung cancer screening

INTERVENTIONS:
Other: lung cancer screening — In the first reading, according to the NCCN lung cancer screening guideline, participants with a solid nodule≤ 5 mm in diameter will be referred to undergo follow-up CT 1 year after the baseline. Participants with a solid nodule 6-14 mm will be referred to undergo follow-up thorax CT 3-6 months after the baseline. Participants with a solid nodule ≥ 15 mm will be referred to a multidisciplinary team for clinical investigation.
  The simulated management will be based on the volume of lung nodule and volume doubling time from the second reading, lung nodules will be reclassified according to the reference values from the European volume-based lung nodule management protocol. According to the European volume-based protocol, the solid and part-solid lung nodules will be reclassified into three groups: nodules with a volume < 100 mm3 (negative), nodules with a volume of 100-300 mm3 (indeterminate), and nodules with a volume > 300 mm3 (positive).

SUMMARY:
European lung cancer screening studies using computed tomography (CT) have shown that a management protocol based on measuring lung nodule volume and volume doubling time (VDT) is more specific for early lung cancer detection than a diameter-based protocol. However, whether this also applies to a Chinese population is unclear. The aim of this study is to compare the diagnostic performance of a volume-based protocol with a diameter-based protocol for lung cancer detection and optimize the nodule management criteria for a Chinese population.

DETAILED DESCRIPTION:
In this population-based study, participants will undergo a low-dose chest CT scan for two rounds. At baseline, the first CT scan will be performed in all participants and their data will be collected. One-year after the baseline, a second CT scan will be performed and data will be collected again. CT images of each participant will be read twice independently by two groups of readers after the baseline and 1-year follow-up scans. In the first reading, the detected lung nodules are evaluated for diameter and managed according to a routine diameter-based protocol. The clinical management of participants are based on the first reading. In the second reading, each scan will be interpreted again by radiologists, blinded to the first reading. Semi-automated volumetry software will be used. The lung nodules will be evaluated for volume and management will be simulated according to a European volume-based protocol. Participants will be followed up and any diagnosis of lung cancer and related information will be collected at the fourth year through the hospital information system and by contacting the participants or their relatives.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-74 years;
* Resident in the Hexi district of Tianjin city for at least 3 years;
* Having no self-reported history of any malignant tumor.

Exclusion Criteria:

* Pregnant woman will be excluded.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
number of clinically diagnosed lung cancer | at the fourth year from baseline
  The number of clinically diagnosed lung cancer will be collected through the hospital information system and by contacting the participants or their relatives using a questionnaire.
number of lung cancer death | at the fourth year from baseline
  The number of lung cancer death will be collected through the hospital information system and by contacting the relatives of the participants using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Ye, Professor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute And Hospital, Tianjin, Tianjin Municipality, China